CLINICAL TRIAL: NCT03295851
Title: Preoperative, Single-dose Intravenous Iron Formulation to Reduce Post-surgical Complications in Patients Undergoing Major Abdominal Surgery: a Pilot Randomised Control Trial (PIRCAS Trial - Pilot)
Brief Title: Preoperative Intravenous Iron Infusion to Reduce Post-surgical Complications: a Pilot Randomised Control Trial
Acronym: PIRCAS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Collaborators: Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FCM001
Record Dates: First submitted 2017-09-19; First posted 2017-09-28 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Anemia; Major Abdominal Surgery; Pre-operative
Keywords: Anemia; Pre-operative; Intravenous Iron; Ferric carboxymaltose; abdominal surgery
MeSH Terms: conditions — Anemia | interventions — ferric carboxymaltose; ferryl iron; ferrous fumarate; Iron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IV Ferric Carboxymaltose (Experimental): Patients in the intervention group will receive preoperative IV ferric carboxymaltose, given as a single dose (15 mg/kg body weight, to a maximum dose of 1000 mg) over 30 minutes.
  Interventions: Drug: Ferric carboxymaltose
- Oral Ferrous Fumarate (Active Comparator): Patients will be given oral iron as per current clinical protocol, which is Ferrous fumarate 200mg twice daily
  Interventions: Drug: Ferrous Fumarate

INTERVENTIONS:
Drug: Ferric carboxymaltose — Patients in the intervention group will receive preoperative IV ferric carboxymaltose, given as a single dose (15 mg/kg body weight, to a maximum dose of 1000 mg) over 30 minutes.
  Other Names: IV Iron
  Arms: IV Ferric Carboxymaltose
Drug: Ferrous Fumarate — Patients will be given oral iron as per current clinical protocol, which is Ferrous fumarate 200mg twice daily.
  Other Names: Oral Iron
  Arms: Oral Ferrous Fumarate

SUMMARY:
Preoperative anemia is common worldwide, ranging from 25% in knee arthroplasties to 60% in colorectal malignancies. In Singapore, about a quarter (27%) of all patients have anaemia prior to operation at a main tertiary center. Currently, the rate of preoperative anemia in Singapore General Hospital (SGH) is 26.6%.

This is an alarming public health issue as the negative impact of preoperative anemia on post-surgical outcomes has been well documented and include increased rates of perioperative blood transfusion, mortality, adverse cardiac and non-cardiac complications including pulmonary complications, wound infections, systemic sepsis and venous thromboembolism, as well as prolonged length of hospital stay and increased healthcare costs. These data suggest that reducing preoperative anemia prior to major surgery is imperative to improve clinical outcomes and decrease healthcare costs.

This study responds to an urgent need to optimize the current standard practice for managing preoperative anemia. It is designed as a randomised, open-label, study to investigate the efficacy of intravenous iron compared to oral iron in patients with anemia undergoing major surgery to reduce surgical complications. To demonstrate the feasibility of conducting such trial in a larger scale, a pilot study with the same design will be conducted. The findings of this pilot study will also inform the study design and sample size for the larger study.

If successful, the results will inform clinical practice guidelines, result in better patient and clinical outcomes, reduce burden on the health care system, and change health-related policy. For example, all forms of intravenous iron therapy are currently not subsidized by the Singapore government which is in stark contrast with allogenic blood transfusion, which is subsidised and readily available at a substantially reduced rate to patients. Hence, it will cost the patients more out of pocket to be treated with intravenous iron than to have allogenic blood transfusion. Incorporating a preoperative anemia correction protocol in the current surgical pathway is a potential strategy to combat healthcare cost inflation and the increasing demand for blood products.

DETAILED DESCRIPTION:
Preoperative anemia is common worldwide, ranging from 25% in knee arthroplasties to 60% in colorectal malignancies. In Singapore, about a quarter (27%) of all patients have anaemia prior to operation at a main tertiary center. Currently, the rate of preoperative anemia in Singapore General Hospital (SGH) is 26.6%.

This is an alarming public health issue as the negative impact of preoperative anemia on post-surgical outcomes has been well documented and include increased rates of perioperative blood transfusion, mortality, adverse cardiac and non-cardiac complications including pulmonary complications, wound infections, systemic sepsis and venous thromboembolism, as well as prolonged length of hospital stay and increased healthcare costs. These data suggest that reducing preoperative anemia prior to major surgery is imperative to improve clinical outcomes and decrease healthcare costs.

This study responds to an urgent need to optimize the current standard practice for managing preoperative anemia. It is designed as an open-label, parallel design pilot randomised control trial to determine the feasibility of conducting a larger scale study powered to investigate reduction in complication rate. There will be two arms, intervention (IV FCM 15mg/kg, up to 1000 mg) and usual care (Ferrous fumarate 200mg twice daily). All participants will be followed for three months from date of operation.

60 participants will be randomly allocated in a 1:1 ratio to either preoperative FCM (intervention) or oral iron (standard care). Participants are stratified to surgical type (upper or lower intestinal surgeries) and surgical approach (laparoscopic or open). The sample size was selected based on the observation that at least 12 participants per group provide adequate measurement precision and power to detect associations. The study aims to balance 15 participants per stratum to account for dropouts and loss to follow up.

Written informed consent will be obtained prior to enrolment in the study. Study data will be entered into a secure data management system and retained for up to 6 years after the study ends, as per institutional guideline. There will be no procedures recorded on electronic media.

The dosing for FCM is based on the maximum dose of intravenous iron that can be safely given in a reasonable time period. The selected dose for the study corresponds with the manufacturer's recommended IV FCM dose for iron repletion in iron deficiency anemia. (Approved product label attached as annex). This dose of 15mg/kg or up to 1000 mg was also the dose used in other similar trials, hence facilitating comparison of results across study populations. As with the manufacturer's recommendation, the drug will be diluted in 250 ml Normal Saline and given over 30 minutes with the patient closely observed for signs and symptoms of hypersensitivity reactions during and for at least 30 minutes following each injection. If contraindication to IV FCM develops, treatment will be stopped and usual care commenced. Such reactions will be recorded and analyzed as an adverse event. The surgeon will be informed of the patient's participation in the study.

The dosing for oral iron would be as per current clinical protocol, which is ferrous fumarate 200mg twice daily.

To determine the effectiveness of a single preoperative dose of IV FCM, compared to oral iron therapy for treating iron deficiency anemia prior to major abdominal surgery, in reducing perioperative blood transfusion requirement and 30-day incidence of postoperative complications. Other secondary objectives:

* To evaluate the effect of intravenous FCM compared with oral iron on change in haemoglobin levels.
* To evaluate the effect of intravenous FCM compared with oral iron on length of hospital stay and mortality.
* To evaluate the effect of intravenous FCM compared with oral iron on health related quality of life.
* To evaluate resource use and costs associated with the treatment with intravenous FCM compared to oral iron.

Reporting of adverse events involves the PI submitting to the approving CIRB the completed SAE Reporting Form within the stipulated timeframe. PI is responsible for informing the institution representative (local SAE resulting in death), sponsor or regulatory bodies as required and appropriate.

Reporting timeline to CIRB:

* SAE that result in death, regardless of causality, should be reported immediately - within 24 hours of the PI becoming aware of the event.
* Local life-threatening (unexpected/ expected) SAE should be reported no later than 7 calendar days after the Investigator is aware of the event, followed by a complete report within 8 additional calendar days.
* Local unexpected SAE that are related events, but not life-threatening, should be reported no later than 15 calendar days after the investigator is aware of the event.
* An increase in the rate of occurrence of local expected SAE, which is judged to be clinically important, should be reported within 15 calendar days after the PI is aware of the event.
* Local expected SAE should be reported annually (together with Study Status Report for annual review).
* Local unexpected and unlikely related SAE that are not life-threatening should also be reported annually (together with Study Status Report for annual review).
* Local unexpected AE that are related events should be reported at least annually (together with Study Status Report for annual review).
* Non-local unexpected SAE that are fatal or life threatening and definitely/probably/possibly related should be reported not later than 30 calendar days after the PI is aware of the event.

All SAEs that are unexpected and related to the study drug will be reported to HSA. All SAEs will be reported to HSA according to the HSA Guidance for Industry "Safety Reporting Requirements for Clinical Drug Trials." The investigator is responsible for informing HSA no later than 15 calendar days after first knowledge that the case qualifies for expedited reporting. Follow-up information will be actively sought and submitted as it becomes available. For fatal or life-threatening cases, HSA will be notified as soon as possible but no later than 7 calendar days after first knowledge that a case qualifies, followed by a complete report within 8 additional calendar days.

The data and safety monitoring will be performed by the Principal Investigator and Co-Investigators, and subjected to audit and monitoring of the practices by Division of Research, SGH as well as CIRB.

The following precautions are in place:

1. Participants with known conditions that might compromise their safety during the administration of the intervention are excluded (see exclusion criteria above)
2. Baseline vitals such as blood pressure, oxygen saturation and heart rate are taken before the commencement of infusion and after the end of infusion
3. The patient is monitored for 30 minutes after the end of IV FCM infusion for any signs and symptoms of hypersensitivity reactions
4. In case of any adverse reactions, participants will be promptly managed according to standard clinical guidelines of adverse events / serious adverse events.

All data will be monitored and reviewed by the PI or Co-investigators. Training will be given to the research coordinator and entry of data from the case report forms for analysis will be verified by a second person from the study team.

Data will be entered on paper, prior to being de-identified and entered electronically for analysis. Existing perioperative surgical, ICU and hospital data will be used to capture patient demographics, procedure urgency, intraoperative procedure and anaesthetic variables, blood product utilisation, mechanical ventilation, delirium/coma, ICU and hospital LOS and major adverse events. Local research staff will enter de-identified study data onto a trial-specific electronic case report form.

Hard copy of research data will be kept in a locked cabinet within the staff-only area of Preoperative Assessment Center, Block 3 Level 1, SGH. Soft copy of all data will be kept on a password protected PC within the hospital's secure network, which is located in the same staff-only area. All data will be de-identified. The participants will not have their NRIC and names displayed in the data. Instead a code will be assigned to each participant to protect the confidentiality of the research data. The key to the code will be kept in a separate access controlled, staff-only office within the department of anesthesiology, SGH. The PI will have access to the identifiers.

For aim 1, the intervention would be deemed feasible if the following three objectives were achieved:

1. 98.5% of subjects to receive study drug within 5 days of enrolment
2. Recruitment of 30 participants within 4 months
3. Complete follow-up in at least 90% of subjects For secondary aims, continuous outcomes, mean differences and 95% CIs will be estimated using analysis of covariance. For binary outcomes risk ratios and risk differences and their 95% CIs will be estimated using binomial regression. For time-to-event outcomes and rates, hazard ratios will be estimated using Cox proportional hazards or negative binomial regression models as appropriate.

The investigator(s)/institution(s) will permit study-related monitoring, audits and/or IRB review and regulatory inspection(s), providing direct access to source data/document.

All data will be monitored and reviewed by the PI or Co-investigators. Training will be given to the research coordinator and entry of data from the case report forms for analysis will be verified by a second person from the study team.

If successful, the results will inform clinical practice guidelines, result in better patient and clinical outcomes, reduce burden on the health care system, and change health-related policy. For example, all forms of intravenous iron therapy are currently not subsidized by the Singapore government which is in stark contrast with allogenic blood transfusion, which is subsidised and readily available at a substantially reduced rate to participants. Hence, it will cost the participants more out of pocket to be treated with intravenous iron than to have allogenic blood transfusion. Incorporating a preoperative anemia correction protocol in the current surgical pathway is a potential strategy to combat healthcare cost inflation and the increasing demand for blood products.

ELIGIBILITY:
Inclusion Criteria:

* Elective major benign or malignant abdominal surgery
* Procedures expected to last 2 hours and/or more OR Anticipated blood loss greater than 500ml
* PAC clinic scheduled before 1 - 4 weeks before surgery
* Male Hb less than 13.0 Gram Per Deciliter OR Female Hb less than 12.0 Gram Per Deciliter
* Diagnosed as having Iron Deficiency: Serum Ferritin level less than 100 Microgram Per Liter OR Serum Ferritin is between less than100 Microgram Per Liter - less than 300 Microgram Per Liter + Transferrin Saturation is less than 20 percent
* Patient is able to receive the infusion 1 - 4 Weeks [at least 7 Days] before the planned operation date.
* Patient is able to provide written, informed consent

Exclusion Criteria:

* Know history of acquired iron overload
* Family history of hemochromatosis or thalassemia or transferrin saturation (TSAT) more than 50 percent
* Treatment with erythropoietin in the previous 12 weeks (3months)
* Known hypersensitivity to Ferric Carboxymaltose or its excipients
* Patients with severe asthma or severe allergy (requiring hospitalization within the last 12 months)
* Pregnancy
* Age less than 21 years
* Inability to communicate or understand study instructions and questionnaire which will be provided in either English, Chinese, Malay or Tamil
* Patient involvement in another Investigational Medicinal Product Trial within the previous 4 weeks prior to randomization that may impact the results of the PIRCAS trial

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-11-22 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the study | four months
  The study can be conducted feasibly at the research site as evidence by:
  1. Number of participants who receive study drug within 5 days of enrollment
  2. Number of participants recruited over 4 months
  3. Number of participants completed the study

SECONDARY OUTCOMES:
effectiveness of a single preoperative dose of IV FCM in treating iron deficiency anemia | one month
  Change in hemoglobin level
the effect of intravenous FCM compared with oral iron on mortality | six month
  all-cause death
the effect of intravenous FCM compared with oral iron on perioperative morbidities | six month
  length of hospital stay
the effect of intravenous FCM compared with oral iron on health related quality of life | three month
  EQ-5D questionnaires
the effect of intravenous FCM compared with oral iron on post operative morbidities | six months
  Postoperative morbidites will be collected using PostOperative Morbidity Survey (POMS) and classified using Clavien-Dindo grading of complications

CONTACTS AND LOCATIONS:
Overall Officials: Hairil Rizal Abdullah, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided